CLINICAL TRIAL: NCT00190931
Title: A Double-Blind Study of Functional Outcomes With Atomoxetine-Hydrochloride and Placebo in Adult Outpatients With DSM-IV Attention-Deficit/Hyperactivity Disorder
Brief Title: A Functional Outcomes Study With Atomoxetine-Hydrochloride and Placebo in Adults With Attention-Deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7066; B4Z-MC-LYBV
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-07-24 (Estimated); Status verified 2006-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride
Drug: placebo

SUMMARY:
The overall primary objective of this study is to test the hypothesis that, compared with placebo,administration of atomoxetine will result in an improved work productivity.

ELIGIBILITY:
Inclusion Criteria:

1. Meet DSM-IV criteria for Attention-Deficit/Hyperactivity Disorder (ADHD).
2. Have a CGI-S-ADHD score of 4 (moderate symptoms) or greater at Visit 1 and Visit 2.
3. Adult Men or Women, 18 years of age or older and not more than 50 years of age at Visit 1.
4. Laboratory results must show no clinically significant abnormalities.
5. Paid employees working 20 hours or more per week and who have been paid in their current place of employment for 6 months or more.

Exclusion Criteria:

1. Meet diagnostic criteria for current major depression, a current anxiety disorder and history of bipolar disorder or any history of a psychotic disorder will be excluded from the study.
2. Are pregnant or are breastfeeding.
3. Have organic brain disease. Have a history of any seizure disorder or patients who have taken or are currently taking anticonvulsants for seizure control.
4. Are taking any psychotropic medication on a regular basis that has central nervous system activity. Must have a washout equal to a minimum of 5 half-lives of that medication prior to Visit 2.
5. Are unstable in any way to participate in this study, in the opinion of the investigator.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400
Dates: Start 2003-11; Study Completion 2005-07

PRIMARY OUTCOMES:
Test the hypothesis that, compared with placebo, administration of atomoxetine for approximately 6 months will result in an improved work productivity,as measured on the Endicott Work Productivity Scale (EWPS) during Study Period II.

SECONDARY OUTCOMES:
To assess the efficacy of atomoxetine in treating core symptoms in adults during Study Period II using the Conners'Adult Attention Deficit/Hyperactivity Disorder Rating Scale-Investigator rated.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Missouri, United States

REFERENCES:
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647